CLINICAL TRIAL: NCT02568163
Title: Influence of Stress on Non Surgical Periodontal Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of subjects were underestimated, which implies a reduction in the number of subjects required.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5502
Record Dates: First submitted 2013-06-25; First posted 2015-10-05 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- questionary (Other)
  Interventions: Other: Non surgical periodontal treatment

INTERVENTIONS:
Other: Non surgical periodontal treatment

SUMMARY:
Treatment of periodontal diseases is influenced by several risk factors. Psychological stress is considered as one of them. Aim of this study is to assess if stress influences results of non surgical periodontal treatment in severe chronic forms of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Severe generalized chronic periodontitis
* Minimum 15 teeth
* Attachment loss > 5mm
* 30% of sites affected- 5% of pockets>5mm
* Bone loss- Bleeding on probing

Exclusion Criteria:

* Patient at risk of endocarditis
* Pregnant women
* Patient under therapy for depression
* Patient treated for periodontal diseases previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Changing depths of periodontal pockets | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de parodontologie, Strasbourg, Bas Rhin, France